CLINICAL TRIAL: NCT02015715
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO6864018 Following Oral Administration in Asian Healthy Subjects
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of RO6864018 in Male, Healthy, Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YP29017
Record Dates: First submitted 2013-11-28; First posted 2013-12-19 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RO6864018 (Experimental): Asian participants will receive a single oral dose of RO6864018 capsule on Day 1. The first dose escalation cohort will receive a single 400 mg oral dose. Dose will be escalated in subsequent cohorts (up to Cohort 4) up to a maximum of 1600 mg, based on safety, pharmacokinetic, and pharmacodynamic data available from lower dose cohorts. The Cohort 5 will include Caucasian participants who will receive a single 1200 mg (or the highest dose well-tolerated by Asian participants, if lower than 1200 mg) oral dose of RO6864018 capsules on Day 1.
  Interventions: Drug: RO6864018
- Placebo (Placebo Comparator): Participants will receive a single oral dose of placebo matching to RO6864018.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO6864018 — A single oral ascending dose of RO6864018 capsules on Day 1.
  Arms: RO6864018
Drug: Placebo — A single oral dose of placebo matching RO6864018 capsules on Day 1.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, single ascending dose study will assess the safety, pharmacokinetics, and pharmacodynamics of RO6864018 in healthy, male, Asian and Caucasian participants. Participants will be enrolled in cohorts and randomized 8:2 to receive a single oral administration of RO6864018 or placebo. Total study duration for each participant is up to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants of ethnic Chinese, Korean, Japanese origin or Caucasian
* No signs of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* Body Mass Index (BMI) between 18 to 30 kilograms per square meter (kg/m^2) inclusive, and a weight range of 50 to 100 kilograms (kg) (110 to 220 pounds [lb]) inclusive at screening
* Non-smokers, or use of less than (<) 10 cigarettes (or equivalent nicotine-containing product) per day

Exclusion Criteria:

* History or symptoms of any significant disease
* Personal or family history of congenital long QT syndrome or sudden death
* Any confirmed significant allergic reactions against any drug, or multiple drug allergies (non-active hay fever is acceptable)
* Positive results for anti-nuclear antibody (ANA), anti-mitochondrial antibody (AMA), anti-smooth muscle antibody (ASMA) and thyroid peroxidase antibody
* Suspicion of regular consumption of drug of abuse
* History (within 3 months of screening) of alcohol consumption exceeding 14 units per week on average (1 unit = 10 grams of alcohol)
* Participants who have received Interferon (IFN) or peginterferon within 8 weeks prior to dosing
* Use of any medication (prescription or over the counter [OTC], including health supplements and herbal remedies) within 2 weeks before the first dose of study medication
* Positive Hepatitis A immunoglobulin M antibody (HAV IgM Ab), Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab) or human immunodeficiency virus antibody (HIV Ab) at screening
* Donation or loss of blood of greater than 500 milliliters (mL) within 90 days prior to dosing
* Have participated in other clinical studies within 60 days prior to study randomization

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Baseline up to Day 29

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of RO6864018 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUC0-inf of Active Metabolite RO6871765 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUC0-inf of Prodrug Metabolite RO6870868 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUC0-inf of Minor Metabolite RO6872373 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Area Under the Plasma Concentration Time Curve From Time Zero to Last Measurable Concentration (AUClast) of RO6864018 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUClast of Active Metabolite RO6871765 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUClast of Prodrug Metabolite RO6870868 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
AUClast of Minor Metabolite RO6872373 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Maximum Observed Plasma Concentration (Cmax) of RO6864018 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Cmax of Active Metabolite RO6871765 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Cmax of Prodrug Metabolite RO6870868 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Cmax of Minor Metabolite RO6872373 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Time to Maximum Plasma Concentration (Tmax) of RO6864018 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Tmax of Active Metabolite RO6871765 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Tmax of Minor Metabolite RO6872373 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
RO6864018 Urine Concentration | Pre-dose (0-4 hours before dosing), 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-Day 1 dose
Active Metabolite RO6871765 Urine Concentration | Pre-dose (0-4 hours before dosing), 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-Day 1 dose
Prodrug Metabolite RO6870868 Urine Concentration | Pre-dose (0-4 hours before dosing), 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-Day 1 dose
Minor Metabolite RO6872373 Urine Concentration | Pre-dose (0-4 hours before dosing), 0-4, 4-8, 8-12, 12-24, 24-36, and 36-48 hours post-Day 1 dose
Apparent Terminal Elimination Half-Life (T1/2) of RO6864018 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
T1/2 of Active Metabolite RO6871765 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
T1/2 of Prodrug Metabolite RO6870868 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
T1/2 of Minor Metabolite RO6872373 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Serum Interferon alpha Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum Interferon-Gamma-Inducible Protein-10 (IP-10) Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum Interleukin (IL)-6 Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum IL-10 Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum IL-12 Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum Neopterin Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Serum p40 (IL-12B) Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Interferon-Stimulated Gene-15 (ISG-15) Messenger Ribonucleic Acid (mRNA) Levels in Whole Blood | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Myxovirus Resistance 1 (MX-1) Gene mRNA Levels in Whole Blood | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Oligoadenylate Synthetase 1 (OAS 1) Gene mRNA Levels in Whole Blood | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Toll-Like Receptor 7 (TLR7) Gene mRNA Levels in Whole Blood | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose
Tmax of Prodrug Metabolite RO6870868 | Pre-dose (0 hour), 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, 36 and 48 hours post-Day 1 dose
Serum Tumor Necrosis Factor Alpha Levels | Pre-dose (0 hours), 3, 6, 12, 18, 24, 36, and 48 hours post-Day 1 dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Singapore (2):
  - Changi General Hospital; Clinical Trial & Research unit, Singapore
  - Singapore